CLINICAL TRIAL: NCT02080455
Title: A Phase 1, Open-Label, Randomized, 2-Arm Study to Evaluate the Effect of Atorvastatin, a Weak CYP3A4 Inhibitor, on the Pharmacokinetics of Lomitapide in Healthy Subjects
Brief Title: Evaluate the Effect of Atorvastatin on the Pharmacokinetics of Lomitapide in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AEGR-733-024
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Effect of Atorvastatin on the Pharmacokinetics of Lomitapide
MeSH Terms: interventions — BMS201038; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lomitapide & Atorvastatin - Taken Together (Experimental): 2 single oral doses of lomitapide (20 mg) with a 14-day washout between (Day 1 & Day 15)
  11 single oral doses of atorvastatin (80 mg) (Day 11 through day 21)
  Interventions: Drug: lomitapide; Drug: Atorvastatin
- Lomitapide & Atorvastatin - Approx. 12 hours between (Experimental): 2 single oral doses of lomitapide (20 mg) with a 14-day washout between (Day 1 & Day 15)
  11 single oral doses of atorvastatin (80 mg) (Day 12 through day 22)
  Interventions: Drug: lomitapide; Drug: Atorvastatin

INTERVENTIONS:
Drug: lomitapide — 20 mg dose
  Other Names: Juxtapid
Drug: Atorvastatin — 80 mg
  Other Names: Lipitor

SUMMARY:
The primary objective of this study is to assess the effect of atorvastatin, a weak cytochrome P450 (CYP) 3A4 inhibitor, on the pharmacokinetics (PK) of lomitapide and its 2 primary metabolites, M1 and M3.

DETAILED DESCRIPTION:
This study will be a single center, randomized, open-label, 2-arm study to evaluate the effects of atorvastatin, a weak CYP3A4 inhibitor, on the PK of lomitapide in healthy male and female subjects when atorvastatin is administered simultaneously with lomitapide and when it is administered 12 hours after lomitapide.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 18 and 55 years of age inclusive
2. BMI between 18.5 and 32.0 kg/m2, inclusive; total body weight of >110 lbs (50 kg);
3. in good health, determined by no clinically significant or relevant abnormalities identified by a detailed medical history and medical exam
4. creatine phosphokinase, AST, and ALT levels must be below 1.5 times the upper limit of normal
5. clinical laboratory evaluations within the reference range for the test laboratory
6. negative test for selected drugs of abuse
7. negative hepatitis panel and negative HIV antibody screens
8. males will either be sterile or agree to use approved methods of contraception
9. all females must have a negative serum beta human chorionic gonadotropin pregnancy test and will be required to use a medically acceptable method of contraception.
10. able to comprehend and willing to sign an Informed Consent Form

Exclusion Criteria:

1. significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, or psychiatric disorder
2. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
3. history of stomach or intestinal surgery or resection
4. history of Gilbert's Syndrome or suspicion of Gilbert's Syndrome
5. subjects who have an abnormality in the 12-lead ECG
6. use of any drugs of abuse for 6 months prior to Check-in;
7. subjects who consume more than 14 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse within 1 year prior to Check-in
8. use of any tobacco- or nicotine-containing products within 6 months prior to Check-in;
9. participation in any other investigational study drug trial within 30 days prior to Check-in;
10. use of any prescription medications/products within 14 days prior to Check-in unless deemed acceptable by the Investigator and Sponsor
11. use of any over-the-counter, nonprescription preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator and Sponsor
12. use of alcohol-, grapefruit- (including star fruit), or caffeine-containing foods or beverages within 72 hours prior to Check-in and through Study Completion
13. poor peripheral venous access;
14. donation of blood (500 mL) from 30 days prior to Screening through Study Completion
15. receipt of blood products within 2 months prior to Check-in;
16. any acute or chronic condition, scheduled hospitalization (inclusive of elective surgery during study) or scheduled travel prior to completion of all study procedures which, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study;
17. subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2014-03-07 (Actual); Study Completion 2014-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sumeray, MD, Study Chair — Cheif Medical Officer; T. Alex King, MD, CPI, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Inc, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lomitapide & Atorvastatin - Taken Together: 2 single oral doses of lomitapide (20 mg) with a 14-day washout between (Day 1 & Day 15)
  11 single oral doses of atorvastatin (80 mg) (Day 11 through day 21)
  lomitapide: 20 mg dose
  Atorvastatin: 80 mg
- Lomitapide & Atorvastatin - Approx. 12 Hours Between: 2 single oral doses of lomitapide (20 mg) with a 14-day washout between (Day 1 & Day 15)
  11 single oral doses of atorvastatin (80 mg) (Day 12 through day 22)
  lomitapide: 20 mg dose
  Atorvastatin: 80 mg
Period: Overall Study
Arm/Group | Lomitapide & Atorvastatin - Taken Together | Lomitapide & Atorvastatin - Approx. 12 Hours Between
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lomitapide & Atorvastatin - Taken Together | Lomitapide & Atorvastatin - Approx. 12 Hours Between | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9.1) | 39 (9.5) | 40 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 12 | 13
  Not Hispanic or Latino | 15 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 8 | 13 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum observed plasma concentration of lomitapide and its 2 primary metabolites (M1 & M3), following administration of lomitapide alone and coadministered with atorvastatin simultaneously (Arm 1)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK of Lomitapide (Lomitapide Alone): PK of lomitapide following administration of lomitapide alone
- PK of Lomitapide (Coadministered Simultaneously): PK of lomitapide following administration of lomitapide coadministered with atorvastatin simultaneously
- PK of M1 (Lomitapide Alone): PK of M1 following administration of lomitapide alone
- PK of M1 (Coadministered Simultaneously): PK of M1 following administration of lomitapide coadministered with atorvastatin simultaneously
- PK of M3 (Lomitapide Alone): PK of M3 following administration of lomitapide alone
- PK of M3 (Coadministered Simultaneously): PK of M3 following administration of lomitapide coadministered with atorvastatin simultaneously
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
ng/mL | 0.940 (34.5) | 2.00 (52.9) | 2.24 (22.8) | 2.11 (31.9) | 32.3 (40.6) | 27.2 (62.0)

2. Primary Outcome: Tmax
Description: Time to reach maximum observed plasma concentration of lomitapide and its 2 primary metabolites (M1 & M3), following administration of lomitapide alone and coadministered with atorvastatin simultaneously (Arm 1)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
hr | 6.00 [3.00 to 10.0] | 10.0 [3.00 to 23.8] | 6.02 [4.00 to 10.0] | 10.0 [4.00 to 23.8] | 4.00 [3.00 to 12.0] | 6.00 [3.00 to 23.8]

3. Primary Outcome: AUC0-t
Description: Area under the concentration-time curve from zero to the last quantifiable concentration of lomitapide and its 2 primary metabolites (M1 & M3), following administration of lomitapide alone and coadministered with atorvastatin simultaneously (Arm 1)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
ng*hr/mL | 36.4 (38.4) | 71.5 (45.3) | 76.8 (34.4) | 76.3 (36.0) | 434 (65.5) | 475 (55.0)

4. Secondary Outcome: Cmax
Description: Maximum observed plasma concentration of lomitapide and its 2 primary metabolites (M1 & M3) following administration of lomitapide alone and coadministered with atorvastatin 12 hours apart (Arm 2)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and have evaluable PK data. 1 subject was removed from formal statistical analysis due to all BLQ values on Day 1 for lomitapide, M1 and M3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK of Lomitapide (Coadministered 12 Hours Apart): PK of lomitapide following administration of lomitapide coadministered with atorvastatin 12 hours apart
- PK of M1 (Coadministered 12 Hours Apart): PK of M1 following administration of lomitapide coadministered with atorvastatin 12 hours apart
- PK of M3 (Coadministered 12 Hours Apart): PK of M3 following administration of lomitapide coadministered with atorvastatin 12 hours apart
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 15 | 16 | 15 | 16 | 15 | 16
ng/mL | 1.09 (49.8) | 1.39 (40.0) | 2.38 (25.5) | 2.66 (25.4) | 28.5 (29.9) | 35.9 (27.3)

5. Primary Outcome: AUC0-∞
Description: Area under the concentration-time curve from zero to infinity of lomitapide and its 2 primary metabolites (M1 & M3), following administration of lomitapide alone and coadministered with atorvastatin simultaneously (Arm 1)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and had evaluable PK data. 2 subjects were removed from formal statistical analysis of "PK of M3 (Lomitapide alone)" due to missing value of AUC0-∞ for Analyte M3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 14 | 16
ng*hr/mL | 40.4 (40.8) | 76.7 (45.1) | 79.1 (34.7) | 78.7 (36.3) | 469 (68.6) | 487 (544)

6. Primary Outcome: t1/2
Description: Apparent terminal elimination half-life of lomitapide and its 2 primary metabolites (M1 & M3), following administration of lomitapide alone and coadministered with atorvastatin simultaneously (Arm 1)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and have evaluable PK data. 2 subjects were removed from formal statistical analysis of "PK of M3 (Lomitapide alone)" due to missing value of AUC0-∞ for Analyte M3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 14 | 16
hr | 50.7 (22.1) | 50.4 (21.8) | 34.0 (17.7) | 35.2 (16.2) | 50.2 (25.6) | 43.2 (18.4)

7. Secondary Outcome: Tmax
Description: Time to reach maximum observed plasma concentration of lomitapide and its 2 primary metabolites (M1 & M3) following administration of lomitapide alone and coadministered with atorvastatin 12 hours apart (Arm 2)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 15 | 16 | 15 | 16 | 15 | 16
hr | 8.02 [4.00 to 12.0] | 8.00 [5.00 to 11.8] | 8.00 [4.00 to 12.0] | 8.00 [5.07 to 11.8] | 6.00 [3.00 to 10.0] | 5.00 [3.00 to 8.00]

8. Secondary Outcome: AUC0-t
Description: Area under the concentration-time curve from zero to the last quantifiable concentration of lomitapide and its 2 primary metabolites (M1 & M3) following administration of lomitapide alone and coadministered with atorvastatin 12 hours apart (Arm 2)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 15 | 16 | 15 | 16 | 15 | 16
ng*hr/mL | 38.8 (40.8) | 50.5 (26.0) | 68.3 (33.0) | 77.6 (27.9) | 410 (32.6) | 542 (31.2)

9. Secondary Outcome: AUC0-∞
Description: Area under the concentration-time curve from zero to infinity of lomitapide and its 2 primary metabolites (M1 & M3) following administration of lomitapide alone and coadministered with atorvastatin 12 hours apart (Arm 2)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK Population consisted of all subjects who received at least one dose of study drug and have evaluable PK data. 3 subjects were removed from formal statistical analysis due to BLQ values on Day 1, missing value of AUC0-∞ on Day 1, and missing value of AUC0-∞ on Day 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- PK of Lomitapide (Coadminister 12 Hours Apart): PK of lomitapide following administration of lomitapide coadministered with atorvastatin 12 hours apart
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadminister 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 15 | 16 | 15 | 16 | 14 | 15
ng*hr/mL | 42.8 (39.6) | 55.8 (25.2) | 70.0 (32.8) | 79.2 (27.8) | 406 (30.8) | 553 (32.4)

10. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life of lomitapide and its 2 primary metabolites (M1 & M3) following administration of lomitapide alone and coadministered with atorvastatin 12 hours apart (Arm 2)
Time Frame: Predose and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 15 | 16 | 15 | 16 | 14 | 15
hr | 52.0 (19.5) | 54.7 (28.5) | 31.2 (24.0) | 32.3 (18.2) | 48.0 (33.4) | 49.7 (21.9)

ADVERSE EVENTS:
Arm/Group | Lomitapide & Atorvastatin - Taken Together | Lomitapide & Atorvastatin - Approx. 12 Hours Between
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/16 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lomitapide & Atorvastatin - Taken Together (N=16) | Lomitapide & Atorvastatin - Approx. 12 Hours Between (N=16)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decreased Appitite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Described in site contract.